CLINICAL TRIAL: NCT02442947
Title: Physiological Examination of Textile Solutions for Stress Reduction When Dressed in Protective Garment and Work Clothes and Under Physical and Heat Stress Conditions
Brief Title: Examination of Textile Solutions for Reducing Physiological Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SHEBA-14-1853-YH-CTIL
Record Dates: First submitted 2015-04-29; First posted 2015-05-13 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Physiological Stress
Keywords: stress when dressed; protective garment; work clothes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Research arm (Experimental): 1. 1 day which will include: physician examination,ECG,anthropometric measurements and Vo2max test.
  2. 6 acclimatization days carried out by a standard protocol including a daily 2 hour effort performed in a climatic chamber, which include walk on a treadmill at 5 Km/h on a 2% incline under heat conditions (40 deg. centigrade & 40% HR) and when dressed in shorts.At the sixth day, the subjects will be dressed in a standard work uniform as a baseline exposure. Core (rectal) and skin temperature and heart rate will be monitored continuously.
  3. 4 experiment days carried out by the following protocol: 2 hour walk on a treadmill (5 Km/h,2% incline) under heavy heat stress conditions (30 deg. centigrade,60% RH) and when dressed each time with different clothing out of 4 options:
     1. NBC protective garment (charcoal base).
     2. combat garment.
     3. 2 different types of work uniforms. physiological stress will be examined based on rectal temperature and heart rate measurements.
  Interventions: Other: clothing type, protective garments of Paul Boye Technologies

INTERVENTIONS:
Other: clothing type, protective garments of Paul Boye Technologies — The experiment aimed at evaluating the physiological stress obtained when dressed in different clothing (NBC protective garment [charcoal base], combat garment and 2 different types of work uniforms- (1)50% cotton and 50% polyester (2)80% cotton and 20% polyester) and during exertion under heat conditions.

SUMMARY:
Using protective or combat garments under heavy heat stress conditions, during rest or exertion, may hinder the body's ability to effectively exchange heat with the environment and thereby can lead to heat injuries. The purpose of this research is to physiologically examine the new textile solutions that are planned to be integrated in the protective garments, combat garments and work uniforms in the army, by evaluating the physiological stress obtained during exertion under hot climatic conditions.

DETAILED DESCRIPTION:
10 young, healthy civilian volunteers will participate in this study. After reading and signing an informed consent form, all subjects will undergo medical examination which includes ECG, anthropometric measurements and Vo2max test. Afterwards, the subjects will perform 6 acclimatization days carried out by the standard protocol of Heat Tolerance Test (HTT). After acclimatization, the subjects will undergo 4 experiment days under heavy heat stress in a climatic chamber, dressed in each experiment day with one out of 4 clothing combinations (NBC protective garment [charcoal base], combat garment and 2 different types of work uniforms). Physiological stress will be evaluated from rectal temperature and heart rate measurements.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-30 years.
* Healthy civilian volunteers.
* Without known medical illness or medication use.

Exclusion Criteria:

* The existence or suspicion of existing cardiac or respiratory disease.
* Hypertension.
* Diabetes.
* Psychiatric condition.
* Any muscles or skeledon condition.
* Any hormonal disease or any other chronic illness that may inhibit participation in the experiment.
* Infectious disease 3 days prior to the experiment.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-06; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
physiological strain (composite) | 10 days for each participant
  The physiological strain will be determined by body core temperature and heart rate of the subjects during a heat tolerance test (HTT).

SECONDARY OUTCOMES:
Rectal temperature | 10 days for each participant
  The rectal temperature will be monitored by a rectal thermistor during each heat tolerance test (HTT).
Skin temperature | 10 days for each participant
  The skin temperature will be monitored by skin thermistors located at 3 sites (chest, arm and leg).
Heart rate | 10 days for each participant
  The heart rate will be monitored using a wearable heart rate monitor (Polar® sensor and heart rate monitor watch).
Sweat rate (composite) | 10 days for each participant
  Sweat rate will be calculated from the patients' body weight and fluid balance.

CONTACTS AND LOCATIONS:
Overall Officials: Ofir Frenkel, M.D, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Tel Litwinsky, Ramat- Gan, Israel